CLINICAL TRIAL: NCT01241175
Title: The Effect of Intravenous Magnesium Sulfate on Intraocular Pressure Following Tracheal Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 4286
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2009-03

CONDITIONS: Increased Intra Ocular Pressure (IOP)
Keywords: IOP; ophthalmic anesthesia; magnesium sulfate
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- magnesium sulfate (Experimental)
  Interventions: Drug: Magnesium Sulfate
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Magnesium Sulfate
  Arms: magnesium sulfate
Drug: normal saline
  Arms: normal saline

SUMMARY:
The aim of this study is to assess the effect of preoperatively administered intra venous magnesium sulfate in attenuating pressure response to laryngoscopy and endotracheal intubation in adult patients scheduled for elective non ocular surgery

ELIGIBILITY:
Inclusion Criteria:

* 18 to 38 years old
* ASA I
* scheduled for elective ENT ambulatory surgeries under general anesthesia

Exclusion Criteria:

* specific major hepatic, renal and cardio-vascular disease
* known to have allergic reaction to magnesium sulphate or other drugs , -hypermagnesemia
* hypocalcemia
* anuria
* heart block
* pregnancy
* any degree of renal insufficiency
* digitalised patients
* positive history of glaucoma or intra ocular hypertension
* refused to participate

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Intra ocular pressure

SECONDARY OUTCOMES:
blood pressure,heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Hilda Mahmoudi, M.D, Study Director — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran